CLINICAL TRIAL: NCT00791609
Title: Evaluation the Feasibility of the FOSTI Device Accurately and in a Real Time Way to Differentiate Malignant From Benign Tissue (Performed ex Vivo) in Cancer Surgery
Brief Title: Evaluation the Feasibility of the FOSTI Device
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Optivasive Ltd. (Industry)
Responsible Party: Anatoliy Babchenko, Optivasive Ltd.
Other Study IDs: OpVe-HI-08-001
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2008-11-14 (Estimated); Status verified 2008-11

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Feasibility of accurate differentiation between malignant and benign tissue using the FOSTI device on surgically removed tissue

DETAILED DESCRIPTION:
Characterization of the optical fiber sensor's interaction with the tissue.

Creating a database of tissue lesions and their 'optical signature' (lesion classifier).

Optimization of the FOSTI device by minimizing the false-positive and false-negative results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of all ages.
* Subject is able, agree and sign the Informed Consent Form.

Exclusion Criteria:

* Subject has any conditions, which precludes compliance with study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of subjects who undergo cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Anatoliy Babchenko, Study Director — Optivasive Ltd.